CLINICAL TRIAL: NCT05899530
Title: Evaluation of Dentoskeletal Changes After Expansion Using Invisalign Versus Conventional Expander Prospective Clinical Study
Brief Title: Dentoskeletal Changes Expansion Using Invisalign Versus Conventional Expander
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amr Samir Abdo Ibrahim, AzharU, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlazharU ASAIbrahim; S.A.Saleh (Registry Identifier: Saleh Anwar Saleh); M.A.Salem (Registry Identifier: Mohamed Ahmad Salem); M.A.Abdarrazik (Registry Identifier: Mohsena Ahmad Abdarrazik)
Record Dates: First submitted 2023-05-25; First posted 2023-06-12 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Expansion of Maxillary Arch; Maxillary Hypoplasia
Keywords: Expander; Hyrax; Invisalign
MeSH Terms: conditions — Retrognathia | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Intervention Model Description: Expansion of maxillary arch by 2 different techniques including conventional expander in one group compared with expansion with clear aligner.
Who Masked: Outcomes Assessor
Masking Description: Invisalign versus conventional expander
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional expander (Active Comparator): Expansion using conventional orthodontic expander(hyrax)
  Interventions: Device: Conventional expander
- Invisalign (Experimental): Expansion with Invisalign appliance
  Interventions: Device: Invisalign

INTERVENTIONS:
Device: Invisalign — Expansion using Invisalign versus conventional expander
  Other Names: Hyrax
  Arms: Invisalign
Device: Conventional expander — conventional expander
  Arms: Conventional expander

SUMMARY:
Cbct evaluation of dentoskeletal changes after expansion using Invisalign versus conventional expander

DETAILED DESCRIPTION:
Using cbct for evaluation of dentoskeletal changes after expansion using Invisalign versus conventional expander hyrax

ELIGIBILITY:
Inclusion Criteria:

* Age (12-16)
* Good oral hygiene
* Constricted maxilla or moderate crowding

Exclusion Criteria:

* Patient receive drugs
* Periodontal diseas
* Past Orthodontic treatment

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-07-22 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Linear amount of midpalatal Suture opening | 4 months
  Apperance of Distema , calculate the amount of general space

CONTACTS AND LOCATIONS:
Overall Officials: Saleh A Saleh, Professor, Study Director — Al-Azhar University; Mohamad A Salem, Professor, Study Director — Al-Azhar University; Mohsena A Abdarrazik, Lecturer, Study Director — Al-Azhar University

IPD SHARING:
Plan to Share IPD: No